CLINICAL TRIAL: NCT05298995
Title: Phase I Study of Anti-GD2 Chimeric Antigen Receptor-Expressing T Cells in Pediatric and Young Adult Patients Affected by Relapsed/Refractory Central Nervous System Tumors
Brief Title: GD2-CAR T Cells for Pediatric Brain Tumours
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Franco Locatelli, Head of the Department of Pediatric Hematology/Oncology and Cell and Gene Therapy, Bambino Gesù Hospital and Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GD2CAR02
Record Dates: First submitted 2022-03-18; First posted 2022-03-28 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Brain Tumor, Pediatric; Medulloblastoma, Childhood; Embryonal Tumor; High Grade Glioma; Diffuse Midline Glioma; Diffuse Intrinsic Pontine Glioma; Brain Tumor Adult
Keywords: Brain tumors; high grade glioma; medulloblastoma; Diffuse Midline Glioma; Diffuse Intrinsic Pontine Glioma; CAR T cell; GD2-antigen; Immunotherapy; Pediatric Central Nervous System tumours; Central nervous system tumour young adults
MeSH Terms: conditions — Brain Neoplasms; Medulloblastoma; Neoplasms, Germ Cell and Embryonal; Glioma; Diffuse Intrinsic Pontine Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ARM A: MB/other embryonal tumor (Experimental): After a lymphodepleting regimen, patients affected by relapsed/refractory MB/other embryonal tumor will receive 1.0 to 6.0 x 10⁶/kg GD2 Chimeric Antigen Receptor (CAR) positive T cells.
  Interventions: Biological: GD2-CART01 (iC9-GD2-CAR T-cells)
- ARM B: Hemispheric HGG (Experimental): After a lymphodepleting regimen, patients affected by relapsed/refractory hemispheric high grade glioma will receive 1.0 to 6.0 x 10⁶/kg GD2 Chimeric Antigen Receptor (CAR) positive T cells.
  Interventions: Biological: GD2-CART01 (iC9-GD2-CAR T-cells)
- ARM C: Thalamic HGG, DMG, DIPG and other rare CNS tumors not included in Arm A and B (Experimental): After a lymphodepleting regimen, patients affected by relapsed/refractory thalamic HGG, DMG, DIPG and other rare CNS tumors not included in Arm A and B will receive 1.0 to 6.0 x 10⁶/kg GD2 Chimeric Antigen Receptor (CAR) positive T cells.
  Interventions: Biological: GD2-CART01 (iC9-GD2-CAR T-cells)

INTERVENTIONS:
Biological: GD2-CART01 (iC9-GD2-CAR T-cells) — Following a lymphodepleting treatment with conventional chemotherapy, patients will be treated with 1.0 to 6.0 x 10⁶/kg GD2 Chimeric Antigen Receptor (CAR) positive T cells, infused i.v. as a single dose

SUMMARY:
The purpose of this study is to test the safety and efficacy of iC9-GD2-CAR T-cells, a third generation (4.1BB-CD28) CAR T cell treatment targeting GD2 in paediatric or young adult patients affected by relapsed/refractory malignant central nervous system (CNS) tumors. In order to improve the safety of the approach, the suicide gene inducible Caspase 9 (iC9) has been included.

DETAILED DESCRIPTION:
The study will consist of a Phase I, dose escalation phase aimed at evaluating the safety and feasibility of intravenous injections of autologous iC9-GD2-CAR T-cells in patients with refractory/relapsed malignant CNS tumors.

Considering the peculiar potential risks associated with the treatment of CNS tumors, the study has been designed to enrol patients in 3 different arms depending on the histology and location of the disease. This model of enrollment is aimed at testing the safety sequentially, starting from categories of patients at lower risk of severe intracranial hypertension first, and subsequently proceeding with patients at proportionally increased risk. In particular, the three arms explored will be relapsed or refractory:

* ARM A: MB/other embryonal tumor
* ARM B: Hemispheric HGG
* ARM C: Thalamic HGG, DMG, DIPG and other rare CNS tumors not included in Arm A and B

Eligible patients will undergo leukapheresis in order to harvest T cells, which will be manufactured to obtain the autologous CAR T product iC9-GD2-CAR T-cells, a GD2-targeting CAR T product. Briefly, the patients will be treated with a lymphodepleting regimen containing conventional chemotherapic agents and subsequently will receive a single infusion of GD2-CART01.

Moreover, the product contains a suicide gene safety switch (namely inducible Caspase 9): in case of relevant toxicities, the patient will receive the dimerizing agent in order to activate the apoptotic pathway in the infused T cells.

After infusion of CAR T cells, the patients will enter a 5-year active follow-up period (for disease follow-up). A conventional 15-year follow-up will be performed as per regulatory requirements in patients receiving gene therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Imaging assessments performed within 14 days of start of treatment
2. Age: 6months-30years
3. Measurable or evaluable disease on at least 2 dimensions on MRI at the time of treatment enrollment
4. Karnofsky/Lansky≥60
5. Recoverfromthetoxiceffectsofpreviousradiationandchemotherapies:grade4and or 3 non-hematologic toxicities must have resolved to grade ≤ 2; in presence of chronic complications (i.e. treatment-associated thrombocytopenia), patient must be clinically stable, according to the opinion of the treating physicians, and meet all other eligibility criteria
6. Positioning of an implantable intraventricular access device (CodmanHolterRickham reservoir, Integra LifeSciences, NJ, U.S.A) and a microdialysis probe (71 high cutoff microdialysis bolt catheter, M Dialysis AB, Stockholm Sweden)
7. Written and signed informed consent from patients, parents or legal guardians. For subjects < 18 year-old their legal guardian must give informed consent. In addition, pediatric subjects will be included in age-appropriate discussion and written informed assent will be obtained for those greater than or equal to 7 years of age, when appropriate
8. Patients of childbearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study and for four months after receiving the preparative regimen
9. Females of childbearing potential must have a negative pregnancy test because of the potentially dangerous effects on the fetus

Exclusion Criteria:

1. Pregnant or lactating women
2. Severe,uncontrolledactiveinfections
3. HIV or active HCV and/or HBV infection
4. Rapidly progressive disease with life expectancy < 6 weeks
5. Historyofgrade3or4hypersensitivitytomurineprotein-containingproducts
6. Hepatic function: inadequate liver function defined as total bilirubin > 4x upper limit of normal (ULN) or transaminase (ALT and AST) > 6 x ULN based on age and laboratory specific normal ranges
7. Renal function: serum creatinine > 3x ULN for age
8. Blood oxygen saturation < 90%
9. Cardiac function: left ventricular ejection fraction lower than 45% by ECHO
10. Marrow function: absolute neutrophils count (ANC) lower than 500/mm3 and/or platelets lower than 20.000 (not reached by transfusion)
11. Congestive heart failure, cardiac arrhythmia, psychiatric illness, or social situations that would limit compliance with study requirements or in the opinion of the principal investigator (PI) would pose an unacceptable risk to the subject. 12.Concurrent or recent prior therapies, before infusion:

    1. If receiving glucocorticoids, patient must be on a stable or weaning dose for at least 7 days prior to infusion. Recent or current use of inhaled/topical/non- absorbable steroids is not exclusionary. Subjects receiving steroid therapy at physiologic replacement doses only are allowed provided there has been no increase in dose for at least 2 weeks prior to starting apheresis
    2. Systemic chemotherapy in the 3 weeks preceding infusion
    3. Immunosuppressive agents less than or equal to 30 days
    4. Radiation therapy must have been completed at least 6 weeks prior to enrollment
    5. Otheranti-neoplasticinvestigationalagentscurrentlyorwithin30dayspriorto start of protocol therapy

13.Patient-derived GD2-CART01 production failure: vitality <80%, CD3+ cells <80%, CD3+ CAR+ cells <20%, CD3+ CAR+ antitumor activity <60% in functional co-culture assay at an Effector: Target ratio 1:1, viable CAR+ cells upon AP1903 exposition >20%, RCR positivity, Vector Copy Number >10, non-sterility, endotoxin contamination (> 1 EU/ml)

Ages: 6 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2038-11 (Estimated)

PRIMARY OUTCOMES:
Safety and definition of the MTD/RD | 4 weeks after CAR T cell infusion
  To evaluate the safety of the infusion of iC9-GD2-CAR-T cells at different escalating/de-escalating doses and establish the dose limiting toxicity (DLT) and the maximum tolerated dose/recommended dose (MTD/RD) of the cellular product

SECONDARY OUTCOMES:
In vivo expansion and persistence | Up to 5 years
  To assess the in vivo persistence and expansion of the infused CAR T-cells in the peripheral blood (PB) and CSF using immunoassays and transgene detection (Droplet PCR), both for the whole population and the specific T cells subsets
Tumor infiltration | Up to 5 years
  To evaluate the tumor infiltration of the infused T cells by immunohistochemistry (IHC), flow cytometry and/or transgene detection (Droplet PCR), whenever the tumor sample is available after the treatment
iC9-GD2-CAR-T cells clearance after AP1903 infusion | Up to 5 years
  To assess the kinetic of iC9-GD2-CAR-T cells clearance after AP1903 infusion
Serum cytokine profiling | Up to 3 months
  To define the serum and CSF cytokine profile and its correlation with CRS in order to identify a possible predictive profile
Time to progression (TTP) | Up to 5 years
  To evaluate the TTP after infusion
Event-free survival (EFS) | Up to 5 years
  To evaluate the EFS after infusion
Overall survival (OS) | Up to 5 years
  To evaluate the OS after infusion
Disease outcome according to the Response assessment in pediatric neuro-oncology (RAPNO) criteria | Up to 5 years
  umor response assessment through the RAPNO criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Pediatrico Bambino Gesù, Roma, Italy, Italy

IPD SHARING:
Plan to Share IPD: No